CLINICAL TRIAL: NCT06591715
Title: Investigation of Biopsychosocial Characteristics of Individuals Diagnosed with Knee Osteoarthritis
Brief Title: Investigation of Biopsychosocial Characteristics of Individuals with Knee Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Aysima Barlak (Other)
Responsible Party: Sponsor-Investigator, Aysima Barlak, PT, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: SBA 24/862
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: osteoarthritis; biopsychosocial; depression; social isolation; pain; sleep; functionality
MeSH Terms: conditions — Osteoarthritis; Depression; Social Isolation; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Home exercise program — The home exercise program routinely given to individuals with knee OA in addition to their medical treatment will consist of exercises routinely used in the BETY innovation.

SUMMARY:
Since pain and depression are observed together in rheumatic diseases, the concept of limitation caused by the disease and health-related quality of life becomes more determinant than radiological joint damage. Sleep problems observed in OA also increase the level of depression findings and difficulty in movement. The chronic nature of the disease includes issues such as pain, fatigue, sleep problems, loss of function, anxiety, depression, and social isolation, together as in other chronic diseases. This complex structure accompanies a picture in which inflammatory processes are triggered.

When the literature is examined, the necessity of evaluation and methods including all these biopsychosocial characteristics of chronic diseases with multifaceted symptoms is emphasized. On the other hand, although it is stated that the common goal of non-pharmacological treatments is to contribute to biopsychosocial improvement in the patient, it is emphasized that evaluations with biopsychosocial content are insufficient. This situation causes the need for scales that provide a holistic assessment of chronic diseases. When the literature, including individuals diagnosed with osteoarthritis, is analyzed, the inadequacy of the studies providing biopsychosocial evaluation draws attention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis according to ACR knee osteoarthritis diagnostic criteria
* Being in stage 2 or 3 according to Kellgren-Lawrence radiological staging criteria
* To be 18 years of age or older
* Being a reader-writer
* Having read and signed the informed consent

Exclusion Criteria:

* History of major psychiatric illness
* Having malignant disease
* Having chronic infectious or other rheumatologic diseases
* Serious knee trauma or surgical operation in the last 6 months
* Having collagen tissue disease
* History of peripheral vascular disease or neuropathy
* Being in stage 4 according to Kellgren Lawrence radiologic staging criteria
* To have received a physiotherapy program for the relevant knee in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-09-09 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive Exercise Therapy Approach (BETY)- Biopsychosocial Questionnaire | 3 mounths
  The BETY Questionnaire was developed on rheumatic patients and was introduced to the literature as a standardized biopsychosocial measurement tool as a result of improving the definitions of recovery from patients with expert opinions and statistical analysis. Scoring of the scale is done using a 5-point Likert system, each item is scored between 0 and 4 points, and a high total score in the scale consisting of a total of 30 items indicates a high biopsychosocial impact.

SECONDARY OUTCOMES:
Health Asessement Questionnaire (HAQ) | 3 mounths
  It is a questionnaire developed in individuals with rheumatoid arthritis and can be used widely and extensively in all rheumatic disease groups and in a wide range of populations including OA. It has 8 subheadings and consists of a total of 20 questions. The sub-headings include dressing, sitting and staying, eating, walking, hygiene, reaching, grasping and activities of daily living. Each answer is scored between 0 and 3 points and the higher the score, the more difficult the activity is.
Hospital Anxiety Depression Scale (HADS) | 3 mounths
  Although the HADS was developed 20 years ago for the clinical measurement of anxiety and depression levels and was originally developed for hospitalized individuals, it now has a wide spectrum of use and can be used in many situations, including healthy people. Seven of the 14 items provide insight into the level of anxiety, while seven include questions about the level of depression. Each question is scored between 0 and 3, with a higher score indicating higher affect. Anxiety and depression sub-parameters are scored separately and a score of 11 and above is considered abnormal.
Short Form - 36 | 3 mounths
  SF-36 scale will be used to determine the level of health status and quality of life of individuals.SF-36 is a patient-oriented assessment scale created in the United States of America that allows for general health screening.Each sub-parameter is scored between 0 and 100 points and a high score indicates good health status.The SF-36 scale has 8 sub-parameters including general health perception, physical function, social function, pain, mental health, role difficulties due to physical causes, role difficulties due to emotional causes and vitality and includes 11 questions with a total of 36 items.
WOMAC Osteoarthritis Index | 3 mounths
  The most commonly used disease-specific questionnaire for the assessment of disease severity in hip or knee OA is the WOMAC questionnaire recommended by the Outcome Measures in Rheumatology Clinical Trials. WOMAC assesses pain, endurance and physical functioning, functional status and stiffness. This scale has gained increasing acceptance in the assessment of OA since its introduction in 1986. The pain subscale includes five items asking about pain with activity, at rest and at night. The stiffness heading includes two questions. The functional status heading includes an assessment of difficulty in 17 different activities. The items are scored from 0 to 4 according to difficulty and the degree of pain and stiffness felt, with a higher total score indicating greater severity of the disease.
Pain Catastrophizing Scale | 3 mounths
  This scale, developed by Sullivan et al. (1995), measures the exaggerated negative mental reaction of individuals to current or anticipated painful experiences and the extent to which they catastrophize pain.The reliability and validity of the Turkish version of the scale was demonstrated by Uğurlu et al. (2017) and consists of 13 items.Each item is scored as never=0, slightly=1, moderately=2, greatly=3 and always=4.A high total score indicates a high degree of catastrophizing of pain.
Tampa Scale of Kinesiophobia | 3 mounths
  This scale is a 17-question scale developed to measure fear of movement/reinjury.The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities
Time Up and Go Test | 3 mounths
  The balance status of the individual is evaluated by getting up from a chair with back support, walking 3 meters at a normal walking speed and returning back to the chair and the time he/she sits on the chair is measured and recorded in seconds.The test is repeated 3 times.
Stair Climb Test | 3 mounths
  In measuring the lower extremity strength and dynamic balance of the individual, the time to ascend and descend 10 steps of 16-20 cm stairs with a handrail as fast as possible is recorded in seconds. The test will be repeated 3 times and the times will be recorded.
30s Sit to Stand test | 3 mounths
  To assess lower limb strength, the subject is asked to stand upright in a chair with arms crossed over the chest and then sit down again. The subject is asked to repeat as quickly as possible for a period of 30 seconds. The score for this assessment test is the number of times the individual stands up fully from a sitting position with arms crossed within 30 seconds.
10 m Walk Tets | 3 mounths
  The individual is asked to walk quickly but without running on a 10-meter path. Three repetitions of the assessment are recorded in seconds.
6 min Walk Test | 3 mounths
  It will be used to assess the functional capacity of the patients. Patients will be asked to walk as long as possible in a 20-meter hospital corridor for 6 minutes in their own rhythm and with standard commands and the distance walked will be recorded in meters.
Muscle Strength | 3 mounths
  Muscle strength will be assessed using the Biodex System 3 Pro® isokinetic device (Biodex Medical Systems Inc., Shirley, NY, USA). Before the first assessment, participants will be recruited to a familiarization session. Each assessment will be preceded by a 10-minute warm-up walk and participants will perform knee flexor and extensor maximal concentric isokinetic muscle strength tests at angular velocities of 180°/s (10 repetitions) and 60°/s (5 repetitions) with a 30-second rest interval. Peak torque (PT) and average power (AP) will be recorded in Newtons (Nm) and watts (W) per meter.
Muscle Endurance | 3 mounths
  In order to evaluate muscular endurance, it will be applied with 20 repetitions at 180°/s angular velocity. A rest period of 30 seconds will be given between the tests. Peak torque measurement will be recorded in Newton meters (Nm). Total work during all repetitions will be recorded in Joules (J).
Proprioception | 3 mounths
  To assess knee proprioception, "active position sense" will be measured at 30°, 45° and 60° by the "Biodex System Pro3 Isokinetic System (Biodex Corp. Shirley NY, USA) as recommended in the literature. Deviation from the target angle will be recorded as absolute angular error, regardless of whether the error is negative or positive. The test will be repeated three times. The mean of the patients' absolute angular errors at each test angle over 3 repetitions will be processed as data

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No